CLINICAL TRIAL: NCT05190562
Title: Effectiveness of Zinc Supplementation in Management of Patients With Symptomatic Benign Migratory Glossitis: A Randomized Control Clinical and Biochemical Study
Brief Title: Effectiveness of Zinc Supplementation in Management of Patients With Symptomatic Benign Migratory Glossitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: mariam hamouda (Other)
Responsible Party: Sponsor-Investigator, mariam hamouda, The Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-RECD-111
Record Dates: First submitted 2021-12-31; First posted 2022-01-13 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Benign Migratory Glossitis
Keywords: Benign Migratory Glossitis; Zinc; Geographic tongue
MeSH Terms: conditions — Glossitis, Benign Migratory | interventions — Zinc Sulfate; Zinc; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zinc Sulphate (Experimental): Zinc Sulphate 25 Mg once daily for one month
  Interventions: Drug: Zinc Sulfate 110 MG (Zinc 25 MG) Oral Tablet

INTERVENTIONS:
Drug: Zinc Sulfate 110 MG (Zinc 25 MG) Oral Tablet — Zinc sulfate is an inorganic compound. It is used as a dietary supplement to treat zinc deficiency and to prevent the condition in those at high risk
  Other Names: Octozinc

SUMMARY:
Effectiveness of Zinc Supplementation in management of patients with symptomatic Benign Migratory Glossitis.

Zinc supplements seems to be a therapeutic option as Migratory glossitis is a chronic disease knowing that it needs no treatment. Zinc deficiency can probably be a causative factor in filiform papillae atrophy. Studies have mentioned the role of zinc in wound healing and maintaining a healthy epithelium, as well as regeneration of filiform papillae. Geographic tongue is a disorder that affects the lingual papillae. It has been shown that zinc sulfate can contribute to the treatment of geographic tongue positively.

DETAILED DESCRIPTION:
Forty-eight patients diagnosed with symptomatic benign migratory glossitis will be selected from Oral Medicine, Periodontology and Oral Diagnosis department, Faculty of dentistry, Ain shams university. Research ethical committee will review the protocol and the procedure will be explained to the patients and they will sign an informed consent.

Seven days after the diagnosis and selection of patients with (BMG), the atrophic areas will be determined and the patients will attend a control checkup in order to exclude those with constant changing patterns of the red atrophic areas with raised keratotic margins. Only those patients who presented with constant atrophic areas with keratotic margins at the control checkup will be included during the study evaluation process, then the selected patient according the following inclusion and exclusion criteria will be randomly allocated into two groups. Patients met the eligibility criteria will be randomly assigned for 2 different groups using computer generated allocation concealment. Group I: Will include 24 patients with symptomatic BMG receiving Zinc Supplementation once daily and zinc rich diet for one month. (study group).Group II: Will include 24 patients with symptomatic BMG receiving zinc rich diet only For one month. (control group). Intensity of the discomfort will be monitored by the patients using the Visual Analogue Scale (VAS). Saliva will be collected from all included patients to evaluate zinc levels before treatment and one month after treatment only.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders are eligible.
2. Adults above 18 years old.
3. Patients who presented at the control checkup with constant atrophic areas with raised keratotic margins.
4. Patients who diagnosed with symptomatic geographic tongue.

Exclusion Criteria:

1. Patients with anemia, oral candidiasis, and indicators for localized irritations (dental caries, affected teeth, sharp teeth edges, dental calculus, faulty dental fillings, and faulty prosthetic procedures).
2. Psoriatic patients.
3. Vulnerable patients (Prisoners, persons with mental disabilities or physical handicaps, children, neonates and pregnant women)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Clinical Score | change from baseline at 8 weeks
  the size of atrophic areas
Subjective Scale | change from baseline at 8 weeks
  intensity of symptoms

SECONDARY OUTCOMES:
Biochemical | change from baseline at 4 weeks
  salivary zinc levels

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Seif Allah, Professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No